CLINICAL TRIAL: NCT01504971
Title: Diagnostic Value of Narrow-band Imaging, Autofluorescence Imaging & White-light Imaging on Gastroesophageal Reflux Disease
Brief Title: Narrow-band Imaging, Autofluorescence Imaging and Gastroesophageal Reflux Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yunsheng Yang, Professor, Department of Gastroenterology and Hepatology, Chinese PLA General Hospital
Other Study IDs: 20111013-001
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux;; Endoscopy;; Esophageal pH monitoring;; Narrow band imaging;; Autofluorescence imaging;; White light imaging;
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastroesophageal reflux disease (GERD)
  Interventions: Other: symptom questionaire; Procedure: pH monitoring; Procedure: Tri-modal imaging endoscopy; Drug: rabeprazole

INTERVENTIONS:
Other: symptom questionaire — GerdQ questionaire
  Other Names: GERD symptom questionaire
Procedure: pH monitoring — 24-hour pH monitoring
  Other Names: Device was from Sierra Company
Procedure: Tri-modal imaging endoscopy — To investigate WLI,NBI and AFI
  Other Names: Device was from Olympus Company
Drug: rabeprazole — 10mg, bid, p.o.
  Other Names: PPI therapy

SUMMARY:
Aim of this study is to compare the efficacy of narrow band imaging (NBI) and autofluorescence imaging (AFI) to distinguish subtle mucosal change related to acid reflux that is not visible in standard white light imaging (WLI) endoscopy, and help indicating the diagnosis of gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
GERD is a common condition that develops when the reflux of gastric and/or duodenal contents causes troublesome symptoms with or without mucosal damage or complications. Despite the high prevalence of GERD in the general population, up to 60% of patients with reflux symptoms is insufficiently characterized as having normal endoscopic finding based on standard WLI endoscopy: non-erosive reflux diseases (NERD).

NBI is an optical-digital imaging technology that uses two specific narrow-banded shot wavelength lights (400-430 nm and 525-555 nm) instead of broad band white light. The NBI contrasts surface structure and vascular architecture of the superficial mucosa and facilitates evaluation of indistinct mucosal morphology. AFI produces real-time computed images of endoscopically detected autofluorescence emitted from endogenous fluorophores in the digestive tract (collagen, nicotinamide, adenine dinucleotide, flavin, and porphyrins) caused by light excitation. The AFI can identify lesions due to differences in tissue fluorescence properties that are not detectable by standard WLI. Hence, our hypothesis is that new endoscopic imaging i.e. NBI and AFI would help to identify subtle mucosal change which indicates the diagnosis of GERD

ELIGIBILITY:
1. Inclusion criteria

   * GERD symptom: heartburn or regurgitation (either one) at least 2 days a week
   * Presence of symptom for longer than 1 month before screening
   * Provision of written informed consent
2. Exclusion criteria:

   * Any known esophageal disease or disorder, other than reflux esophagitis
   * Active or healing gastroduodenal ulcer (except scars)
   * History of esophageal or gastric surgery.
   * Clinically significant heart, lung, liver or kidney disease
   * Allergy to proton-pump inhibitor
   * Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presented with reflux symptoms in outpatient clinic of a general hospital.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhang Li, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Outpatient Department Building, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Fock KM, Teo EK, Ang TL, Tan JY, Law NM. The utility of narrow band imaging in improving the endoscopic diagnosis of gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2009 Jan;7(1):54-9. doi: 10.1016/j.cgh.2008.08.030. Epub 2008 Sep 3. PMID 18852068

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gastroesophageal Reflux Disease (GERD)
Started | 95
Completed | 82
Not Completed | 13
Not completed — Physician Decision | 13

BASELINE CHARACTERISTICS:
Arm/Group | Gastroesophageal Reflux Disease (GERD)
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 52
Region of Enrollment [Number; unit: participants]
  China | 95

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Ability of Each Endoscopic Finding for GERD Symptom.
Description: Patients with GERD symptom receive endoscopic tri-modal imaging within 1 month
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participants: Diagnostic capabilities of White-light Imaging on Gastroesophageal Reflux Disease
- Participants Same to arm1: Diagnostic capabilities of Autofluorescence Imaging on Gastroesophageal Reflux Disease
- Participants Same to Previous Arm: Diagnostic capabilities of GerdQ in the diagnosis of GERD
Arm/Group | Participants | Participants Same to arm1 | Participants Same to Previous Arm
Number analyzed (Participants) | 82 | 82 | 82
percentage of participants | 21 [9 to 32] | 77 [65 to 89] | 60 [45 to 74]

2. Secondary Outcome: Association of Each Endoscopic Finding With Symptom Score
Description: Symptom score is assessed by a self-reported questionnaire
Time Frame: 1 month
Reporting Status: Not Posted

3. Secondary Outcome: Association of Each Endoscopic Finding With pH Monitoring Result
Time Frame: 1 month
Reporting Status: Not Posted

4. Secondary Outcome: Association of Each Endoscopic Finding With Treatment Effect of PPI
Description: Treatment effect of PPI is assessed by changes of symptom score
Time Frame: 2 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Participants: Diagnostic capabilities of WLI in the diagnosis of GERD
- Participants Same to arm1: Diagnostic capabilities of AFI in the diagnosis of GERD
Arm/Group | Participants | Participants Same to arm1 | Participants Same to Previous Arm
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No